CLINICAL TRIAL: NCT06104969
Title: Predictive and Diagnostic Biomarkers for Diabetic Foot Ulcers: Open Wound Master Study
Brief Title: DFC 004 Biomarkers for Active Diabetic Foot Ulcers
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Cathie Spino, ScD, Professor, University of Michigan
Other Study IDs: HUM00231478
Record Dates: First submitted 2023-07-19; First posted 2023-10-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Diabetes
Keywords: diabetic foot ulcer; Diabetic Foot Consortium
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Data collected for this study will be analyzed and stored at the DFC DCC at the University of Michigan. After the study is completed, the de-identified, archived data will be transmitted to and stored at the NIDDK Data Repository, for use by other researchers including those outside of the study.
  With the participant's approval and as approved by the central and local Institutional Review Boards (IRBs), de-identified biological samples will be stored at the DFC Central Laboratory for studies approved by the DFC Steering Committee and eventually in NIDDK Central Repository. Permission for depositing the biological samples in these repositories will be included in the informed consent. The NIDDK Central Repository will also be provided with a code-link that will allow linking the biological specimens with the phenotypic data from each participant, maintaining the blinding of the identity of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic Foot Ulcer: Adult individuals with at least one diabetic foot ulcer who meet inclusion/exclusion criteria

SUMMARY:
This study is a platform study designed to efficiently test multiple biomarkers to identify diabetic foot ulcers (DFUs) with a higher potential for healing versus not healing that ultimately could be applied at the point of care to drive personalized management decisions, and to better inform clinical trials of wound healing interventions

DETAILED DESCRIPTION:
This study is a platform study designed to efficiently test multiple biomarkers to identify diabetic foot ulcers (DFUs) with a higher potential for healing versus not healing that ultimately could be applied at the point of care to drive personalized management decisions, and to better inform clinical trials of wound healing interventions The platform study is designed to be flexible so that it is suitable for a wide range of studies relevant to patients with open (active) DFUs.

This platform study will enroll patients with DFUs seen in an outpatient setting in diabetic foot and wound care clinics across a range of healthcare systems, including community settings and tertiary care hospitals, participating in the DFC.

The platform study will include common procedures that are applicable across the entire spectrum of DFUs (e.g., uniform biospecimen collections, clinical and usual care characteristics, social determinants of health, and patient reported outcomes). Blood, wound fluid (by a variety of methods), wound dressings, and debridement tissue (if debridement is performed during the participant's clinical wound care) will be collected from all participants to support a biorepository for concurrent and future research. Urine samples will be collected if participants agree to provide them, and collection will be encouraged. Biomarker-specific studies requiring additional data or biospecimens not required in the platform study will be included as appendices, as needed. Other biomarker-specific studies that use platform study biospecimens and study data will follow the DFC ancillary study process.

Eligible participants enrolled in the master protocol who signed the informed consent may be enrolled in multiple biomarkers sub studies associated with the master protocol without the need to sign an additional informed consent.

This platform study is non-interventional; no study prescribed agents or therapies are administered.

Eligible and consented participants are managed at each DFC site according to the usual clinical care, which is expected to be in line with the current standards of care recommendations1-3. The study will collect relevant details regarding the care provided at each clinic visit and participant outcomes.

Follow-up for participants will vary based upon the occurrence and timing of healing:

* All participants will be followed every other week for one month and monthly thereafter until the wound is healed or week 52 if the wound has not healed.
* Participants who experience wound healing prior to week 52 will have a confirmation visit 2 weeks later. These participants will also be assessed for recurrence of their DFU at weeks 52 and 78 via phone call or video visit.
* Participants who experience wound healing at week 52 will have a confirmation visit 2 weeks later. These participants will also be assessed for recurrence of their DFU at week 78 via phone call or video visit.
* Participants who do not experience wound healing by week 52 will have an additional phone call or video visit scheduled at week 78 to assess patient-reported wound healing, infection, or amputation with confirmation by electronic medical records (EMR), if available.

Study visits may occur in conjunction with the participant's scheduled clinical follow-up visits. After wound healing has been confirmed, the visit may be conducted by remote means.

The master protocol will enable evaluation of the time to healing over a 78-week period and of expectations on the natural history of wound healing in contemporary DFU participants. It also enables exploring rates of DFU recurrence in those who healed. These data will lead to more accurate DFU-specific standards of care guidelines that will have a direct impact and benefit in the clinical care, for a personalized approach.

General and biomarker-specific analyses will be performed. Participants who share common demographic or clinical characteristics may be pooled across substudies.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Age 18 years or older.
3. Clinically diagnosed with diabetes or meeting the American Diabetes Association (ADA) criteria. [ADA Standards of Clinical Care Diabetes Care 2022, Suppl 1]
4. Open foot ulcer, defined as an open wound from malleolus down. This includes post-surgical wounds within this area left open to heal by secondary intention. In case of multiple ulcers, the largest ulcer will be considered the study index DFU.
5. Agreement to adhere to protocol visits and provide all required biospecimens and clinical data.

Exclusion Criteria:

1. Participation in an interventional clinical trial for DFU within 1 month of Visit 1.
2. Currently receiving radiation to target area or chemotherapy.
3. Gangrene in any portion of the foot with the index ulcer.
4. Planned revascularization or under evaluation for revascularization of the index limb for advanced ischemia within next 4 weeks of Week 0.
5. Severe limb ischemia (SVS WIfl Ischemia grade 3).
6. Any concomitant medical or psychiatric condition that, in the opinion of the investigator(s), would compromise the participant's ability to safely complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diabetes with at least one open diabetic foot ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 52 Weeks
  Proportion of participants with complete wound healing by week 52, defined as complete wound closure where there is skin re-epithelialization without drainage or dressing requirements at two consecutive study visits 2 weeks apart.
DFU Infections | 52 Weeks
  Proportion of participants who develop infections of the index DFU among those with no infections at baseline.
Amputations | 52 Weeks
  Proportion of participants who have an amputation of the limb associated with the index DFU.
Prediction Performance | 52 Weeks
  Measures of prediction performance (e.g., predictive power, AUC, ROC, Akaike information criterion) of biomarker(s) for each of the clinical outcomes: Wound Healing, DFU Infections, and Amputations described above.
  Prediction performance is measured by multiple statistical measures to assess ability of the biomarker to predict event risk for each of the three clinical outcomes.
Biospecimens Count | 52 Weeks
  Proportion of eligible participants providing biospecimens by site, and by type (serum, plasma, wound fluid, wound dressings, wound debridement tissue, urine).
Biospecimen Quality | 52 Weeks
  Proportion of biospecimens of adequate quality by type.
Standard of Care Prescription by Site | 52 Weeks
  Proportion of sites that prescribe the most current SOC into usual care, specifically for: (a) offloading; (b) vascular assessment; and (c) debridement.
Standard of Care Adherence | 52 Weeks
  Proportion of participants who adhere to physician-prescribed SOC therapies for their DFU care.

SECONDARY OUTCOMES:
Time to Healing | Up to 52 Weeks
  Time to healing, defined as the time (in weeks) from baseline to complete healing.
Change from baseline to later of Week 52 or Confirmation Visit in SF-12 Physical Domain Score | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  SF-12 physical domain score.
  SF-12 for physical
  * Score range from 0-100
  * Higher scores indicate better physical health.
Change from baseline to later of Week 52 or Confirmation Visit in SF-12 Mental Domain Score | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  SF-12 mental domain score.
  * Score range from 0-100
  * Higher scores indicate better mental health.
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF subscale leisure score. | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF physical health subscale score. | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF dependence/daily life subscale score. | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF negative emotions subscale score. | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF worried about ulcers/feet subscale score | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in DFS-SF bother by ulcer care subscale score. | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  DFS-SF subscale scores (leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, bother by ulcer care).
  DFS-SF subscale scoring
  * Five-point scale: 1=never to 5=all the time
  * Score is based on sum of all items
  * Scored 0-100 - higher scores indicate better QOL
Change from baseline to later of Week 52 or Confirmation Visit in PROMIS Sleep Disturbance | 52 Weeks
  Change from baseline to later of Week 52 or Confirmation Visit in:
  PROMIS Sleep disturbance.
  * Each items has a 5-point response scale
  * 1=never, 2=rarely, 3=sometimes, 4=often, 5=always
  * Score ranges from 8-40; higher scores indicate greater severity of sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Arizona College of Medicine, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Northwell Health, Lake Success, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No